CLINICAL TRIAL: NCT06421025
Title: Evaluation of Blood Viscosity and Hyperviscosity-related Complications Relationship in Patients With Patients With Polycythemia
Brief Title: Blood Viscosity in Polycythemia Patients
Acronym: POLYVISCO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0915; 2023-A02208-37 (Other: ID-RCB)
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Polycythemia Secondary; Polycythemia, Primary
Keywords: Polycythemia; viscosity; thromboelastometry; thrombosis
MeSH Terms: conditions — Polycythemia Vera; Polycythemia; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with polycythemia: Patients with polycythemia defined as hematocrit level greater than or equal to 49% in men and 48% in women, whatever the suspected etiology. Primitive and secondary polycythemia are eligible in this observational study. Patients should not have start any cytoreductive therapy prior inclusion.

SUMMARY:
Polycythemia (PG) corresponds to an increase in erythrocyte parameters on a blood test. A distinction is usually made between primary and secondary PG. The most common primary PG is Vaquez's disease, a hematological cancer. In Vaquez disease, an increase in hematocrit has been reported to be associated with a logarithmic increase in blood viscosity.

The main complications of primary PGs (especially in Vaquez disease) are thromboembolic complications. In contrast, thromboembolic complications are rarer in secondary PG. In Vaquez disease, a hematocrit ≤ 45% has been defined as the therapeutic goal for significantly reducing thromboembolic risk. However, this has not been established for secondary PGs. All in all, the definition of the 45% threshold is based solely on clinical studies with no obvious biological argument. What's more, simply lowering blood mass through cytoreduction alone does not appear to be sufficient to significantly reduce thromboembolic risk.

To investigator knowledge, there are no studies prospectively evaluating blood viscosity, its determinants and coagulation in different types of polycythemia. Nor are there any data on the direct effect on blood viscosity of the various treatments usually offered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Followed for a diagnosis or suspicion of polycythemia (hematocrit greater than or equal to 49% in men and 48% in women), whatever the suspected etiology.
* Patient affiliated to a social security scheme or similar

Exclusion Criteria:

* Patient having undergone therapeutic bloodletting within 3 months prior to inclusion, or having initiated cytoreductive therapy prior to inclusion.
* Any disease or condition other than polycythemia, chronic or not, likely to induce a change in blood viscosity (at the investigator's discretion)
* Patient participating in another interventional research protocol that may interfere with the present protocol (at the investigator's discretion).
* Patient under guardianship, curatorship or safeguard of justice
* Person under psychiatric care
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polycythemia defined as hematocrit level greater than or equal to 49% in men and 48% in women, whatever the suspected etiology. Primitive and secondary polycythemia are eligible in this observational study. Patients should not have start any cytoreductive therapy prior inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2031-09-10 (Estimated); Study Completion 2031-09-10 (Estimated)

PRIMARY OUTCOMES:
Whole blood viscosity levels in patients with polycythemia | Baseline
  The investigators expect higher blood viscosity values in polyglobulic patients with symptoms of clinical hyperviscosity than in polyglobulic patients without symptoms of clinical hyperviscosity, but no differences in hematocrit between the two polycythemia groups

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie, Hôpital Lyon Sud, Pierre-Bénite, Lyon, France

REFERENCES:
- [Background] Marchioli R, Finazzi G, Specchia G, Cacciola R, Cavazzina R, Cilloni D, De Stefano V, Elli E, Iurlo A, Latagliata R, Lunghi F, Lunghi M, Marfisi RM, Musto P, Masciulli A, Musolino C, Cascavilla N, Quarta G, Randi ML, Rapezzi D, Ruggeri M, Rumi E, Scortechini AR, Santini S, Scarano M, Siragusa S, Spadea A, Tieghi A, Angelucci E, Visani G, Vannucchi AM, Barbui T; CYTO-PV Collaborative Group. Cardiovascular events and intensity of treatment in polycythemia vera. N Engl J Med. 2013 Jan 3;368(1):22-33. doi: 10.1056/NEJMoa1208500. Epub 2012 Dec 8. PMID 23216616
- [Background] Vogel J, Kiessling I, Heinicke K, Stallmach T, Ossent P, Vogel O, Aulmann M, Frietsch T, Schmid-Schonbein H, Kuschinsky W, Gassmann M. Transgenic mice overexpressing erythropoietin adapt to excessive erythrocytosis by regulating blood viscosity. Blood. 2003 Sep 15;102(6):2278-84. doi: 10.1182/blood-2003-01-0283. Epub 2003 May 15. PMID 12750170
- [Background] Wade JP, du Boulay GH, Marshall J, Pearson TC, Russell RW, Shirley JA, Symon L, Wetherley-Mein G, Zilkha E. Cerebral blood flow, haematocrit and viscosity in subjects with a high oxygen affinity haemoglobin variant. Acta Neurol Scand. 1980 Apr;61(4):210-5. doi: 10.1111/j.1600-0404.1980.tb01485.x. PMID 7376820
- [Background] Barbui T, De Stefano V, Ghirardi A, Masciulli A, Finazzi G, Vannucchi AM. Different effect of hydroxyurea and phlebotomy on prevention of arterial and venous thrombosis in Polycythemia Vera. Blood Cancer J. 2018 Nov 26;8(12):124. doi: 10.1038/s41408-018-0161-9. No abstract available. PMID 30478311
- [Result] Pearson TC. Hemorheology in the erythrocytoses. Mt Sinai J Med. 2001 May;68(3):182-91. PMID 11373690